CLINICAL TRIAL: NCT06458517
Title: Pilot Observational Study of Transcutaneous and Intraoral Photobiomodulation in the Prevention and Treatment of Radiomucositis in Head and Neck Cancers Treated by Radiotherapy - RADIO-PBM Trial
Brief Title: Evaluation of Two Methods of Administration of Photobiomodulation in the Context of the Prevention and Treatment of Mucositis Induced by Radiotherapy, During the Treatment of Head and Neck Cancers
Acronym: RADIO-PBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-018
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Neoplasms
Keywords: Radiotherapy; Chemotherapy; Photobiomodulation therapy; Low-level laser therapy; Oral mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral PBM (Other)
  Interventions: Device: Photobiomodulation session - intraoral
- Transcutaneous PBM (Other)
  Interventions: Device: Photobiomodulation session - transcutaneous

INTERVENTIONS:
Device: Photobiomodulation session - intraoral — use of CareMin650TM lightbox(NeoMedLight) in preventive and in case of occurence of grade 1 oral mucositis, in curative purpose
  Arms: Intraoral PBM
Device: Photobiomodulation session - transcutaneous — use of ATP38® phototherapy device (Swiss Bio Inov Europe) in preventive and in case of occurence of grade 1 oral mucositis, in curative purpose
  Arms: Transcutaneous PBM

SUMMARY:
The aim of this feasibility, prospective, single-center trial is to compare an intra-oral Photobiomodulation (PBM) via the Caremin650TM device (NeoMedLight) and a transcutaneous PBM via the ATP 38® device (Swiss Bio Innov) in patients treated with radiotherapy or chemoradiotherapy for cancer of the oropharynx or oral cavity. PBM session will be carried out first at the rate of two sessions per week for preventive purposes, and then, in case of occurence of grade 1 mucositis, three sessions per week with curative purpose.

DETAILED DESCRIPTION:
Oral mucositis (OM) is defined as damage to the mucosa of the oral cavity; it can be due to chemotherapy or radiotherapy. The incidence of OM is 59 to 100% according to studies in patients with oral cavity or oropharyngeal cancer receiving radiotherapy.

Clinically, OM is characterized by erythematous changes in the mucosa, which can progress to oral ulcerations. It can significantly alter the quality of life, the ability to eat, cause weight loss in patients and interfere with the proper realization of anti-tumoral treatment. Additionally, OM may increase the risk of bacteremia and sepsis in immunocompromised patients.

So far, effective management strategies for OM and associated pain are still insufficient. A wide variety of topical and oral agents are available, but effectiveness is still lacking.

Photobiomodulation (PBM) therapy involves the application of visible or infrared light produced by laser diodes or light-emitting diodes (LEDs) to stimulate wound healing, reduce inflammation, and decrease pain.

PBM can be performed in two main ways: intraoral and transcutaneous. Intraoral PBM involves applying red or near-infrared light directly in contact with the oral mucosa, while transcutaneous PBM involves the application of infrared radiation to the skin. Both techniques have shown their effectiveness. Numerous trials have evaluated the impact of PBM in radiomucositis but its use in clinical practice is to date not widespread and heterogeneous.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years old and older);
* Patients with oral cavity or oropharynx cancer treated with radiotherapy or chemo-radiotherapy;
* Karnofsky Performance Status > 60%;
* Able to understand French;
* With signed informed consent;
* Affiliated to French Health Security Insurance

Exclusion Criteria:

* Allergy to polyurethanes;
* Head and Neck tumors that are localized to other sites than oral cavity or oropharynx
* Previous irradiation of Head and Neck (whatever the time lapse between the two irradiations)
* Pregnant and breastfeeding woman;
* Patients with pacemaker device
* Epileptic patients;
* Concomitant treatment or treatment within the 7 days before inclusion with one of several drugs from the following list: fluoroquinolones, cycline, methotrexate, auranofin
* Patients with ophthalmic diseases (such as maculopathy, retinopathy, glaucoma and cataract, retinal damage)
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of oral mucositis (grade ≥ 2) in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Oral mucositis will be graded according to NCI-CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Radiotherapy treatment interruption in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Number of cancelled radiotherapy sessions in comparison to initial treatment plan
Duration of oral mucositis in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Number of days
Number of hospitals stays in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Number of unscheduled hospitalizations
Number of introductions of parenteral nutrition in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Number of days from radiotherapy initiation until artificial nutrition introduction
Infection rate in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Infections graded according to NCI-CTCAE V5.0 criteria
Food intake in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Measured on a weekly basis with the Simple Evaluation of Food Intake (SEFI) tool
Pain level in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Measured with a visual analogic scale (VAS), graded from 0 to 10
Quality of life of patients in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Questionnaire from EORTC: QLQ-C30 with organ specific QLQ-HN35 module
Dry mouth rate in both group (intraoral and transcutaneous PBM) | Until OM resolution, up to 12 weeks
  Graded according to NCI-CTCAE V5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jordan EBER, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Derived] Eber J, Schohn A, Carinato H, Brahimi Y, Schmitt M, Noel G. A Pilot Study Comparing Intraoral and Transcutaneous Photobiomodulation for Oral Mucositis in Head and Neck Cancer Patients Undergoing Radiotherapy or Chemoradiotherapy. J Clin Med. 2025 Apr 2;14(7):2430. doi: 10.3390/jcm14072430. PMID 40217880